CLINICAL TRIAL: NCT03163602
Title: Surgical Treatment of Peri-implantitis. A Randomised Controlled Trial.
Brief Title: Surgical Treatment of Peri-implantitis
Acronym: STP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Principal Investigator, Lisa Heitz-Mayfield, Adj Professor, The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-116
Record Dates: First submitted 2017-04-14; First posted 2017-05-23 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis; Infection; Bone substitutes
MeSH Terms: conditions — Peri-Implantitis; Infections | interventions — Control Groups; Debridement

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group 1 (Active Comparator): Access flap, implant surface decontamination (saline), systemic antibiotics (amoxicillin 500 mg and metronidazole 400 g, 3 x day for 7 days)
  Interventions: Drug: Control group
- Test Group 2 (Active Comparator): Access flap, implant surface debridement, systemic antibiotics (amoxicillin 500 mg, metronidazole 400 g, 3 x day for 7 days), bovine bone substitute material (BioOss®) and collagen membrane (BioGide®)
  Interventions: Device: Test group

INTERVENTIONS:
Drug: Control group — Access flap and debridement
  Other Names: Access flap and debridement
  Arms: Control Group 1
Device: Test group — Regenerative treatment
  Other Names: BioOss®, BioGide® collagen membrane
  Arms: Test Group 2

SUMMARY:
The aim of this randomized controlled study is to evaluate the outcome of surgical treatment of peri-implantitis with and without the use of a bone substitute graft covered by a collagen membrane. There will be a follow up period of 12 months. Outcome measures will include assessments of inflammation, probing depth, recession, radiological parameters and PROMs.

DETAILED DESCRIPTION:
The aim of this randomized controlled study is to evaluate the possible benefit of a regenerative treatment protocol (placing a bone substitute covered by a bioresorbable collagen membrane) compared to surgical treatment alone, for peri-implantitis therapy.

The hypothesis is that there will be a greater number of patients with successful treatment of peri-implantitis following the use of a bone substitute/collagen membrane compared to surgical peri-implantitis therapy without the bone substitute/collagen membrane.

The project will be conducted as a two-armed randomized controlled clinical trial of 1-year duration. Forty systemically healthy patients with ≥1 implant diagnosed with peri-implantitis requiring surgical therapy will be enrolled.

Baseline measurements will be performed after non-surgical therapy (removal supramucosal biofilm/calculus, oral hygiene instruction and correction of prosthetic factors) and treatment of periodontitis.

Baseline measurements will include probing depth, position of mucosal margin, presence of plaque, presence of bleeding and/or suppuration on probing, PROMs and radiographs. Measurements will be recorded at 4 sites per implant.

Following the baseline measurements participants will be randomly assigned to either Control Group (Group 1): access flap and implant cleaning or Test Group (Group 2): access flap, implant cleaning and addition of a bone substitute material covered by a collagen membrane.

Participants in both treatment groups will be prescribed systemic antimicrobials (Amoxicillin 500 mg tds and Metronidazole 400 mg tds) for 7 days starting from the day of surgery.

In addition an antibacterial mouthrinse (chlorhexidine digluconate 0.2%) will be prescribed for a period of 4 weeks following surgery.

Participants will be asked to attend follow-up visits for review of healing (week 1 and 4) and maintenance care (3, 6, 9, and 12 months).

Clinical examinations will be performed by a calibrated blinded examiner at baseline and 12 months after therapy. Clinical measurements will be taken using a periodontal probe at 4 sites per implant to record presence of plaque, bleeding, probing depth and recession of the soft tissue.

PROMS will be assessed at 1 week, 4 weeks and at 12 months. Radiographic assessments Intra-oral radiographs and cone beam CT scan will be obtained prior to surgery and at 12 months. Oral-maxillofacial radiologists will. perform the radiographic analysis and will be blinded to the treatment procedure.

Primary outcome variables include (1) resolution of peri-implantitis (probing depth reduction and absence of BoP, suppuration) (2) recurrence of disease (BoP, suppuration and increase in PPD and progression of bone loss.

ELIGIBILITY:
Inclusion Criteria:

Presence of ≥ 1 implant with a probing depth (PD) ≥ 5 mm with bleeding and/or suppuration (SUP) on probing, and peri-implant bone loss ≥ 3mm with an intraosseous defect component

Exclusion Criteria:

* Smokers > 10 cigarettes per day
* Patients with uncontrolled diabetes mellitus
* Pregnant or lactating women (self reported)
* Patients with a systemic illness that preclude them from oral surgery
* Patients with an allergy to amoxicillin or metronidazole or chlorhexidine.
* Patients requiring antibiotic prophylaxis and Patients who have taken antibiotics in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Composite Success Outcome | 12 months
  Number of participants with treated implant with successful outcome: no bleeding or suppuration on probing, no further bone loss, PD ≤ 5 mm

SECONDARY OUTCOMES:
probing depth change | 12 months
  mm
radiographic bone level change | 12 months
  mm
change in peri-implant soft tissue level | 12 months
  mm
patient reported outcomes | 1, 6, 12 months
  VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Heitz-Mayfield, OdontDr, Principal Investigator — The University of Western Australia
Locations (1):
- The University of Western Australia, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esposito M, Grusovin MG, Worthington HV. Treatment of peri-implantitis: what interventions are effective? A Cochrane systematic review. Eur J Oral Implantol. 2012;5 Suppl:S21-41. PMID 22834392
- [Background] Heitz-Mayfield LJ, Mombelli A. The therapy of peri-implantitis: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:325-45. doi: 10.11607/jomi.2014suppl.g5.3. PMID 24660207
- [Background] Carcuac O, Derks J, Charalampakis G, Abrahamsson I, Wennstrom J, Berglundh T. Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. J Dent Res. 2016 Jan;95(1):50-7. doi: 10.1177/0022034515601961. Epub 2015 Aug 18. PMID 26285807
- [Background] Heitz-Mayfield LJA, Salvi GE, Mombelli A, Loup PJ, Heitz F, Kruger E, Lang NP. Supportive peri-implant therapy following anti-infective surgical peri-implantitis treatment: 5-year survival and success. Clin Oral Implants Res. 2018 Jan;29(1):1-6. doi: 10.1111/clr.12910. Epub 2016 Jun 23. PMID 27335316
- [Derived] Heitz-Mayfield LJA, Heitz F, Koong B, Huang T, Chivers P. Surgical peri-implantitis treatment with and without guided bone regeneration. A randomized controlled trial. Clin Oral Implants Res. 2023 Sep;34(9):892-910. doi: 10.1111/clr.14116. Epub 2023 Jun 29. PMID 37382408